CLINICAL TRIAL: NCT02814994
Title: Respiratory System Compliance Guided Tidal Volume in Moderate to Severe ARDS Patients: A Multicenter Randomized Controlled Study
Brief Title: Respiratory System Compliance Guided VT in Moderate to Severe ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, physician, Zhongda Hospital, Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARDS protocol treatment
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Mechanical Ventilation; ARDS; Ventilator Strategy; Outcome
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tidal volume guided by respiratory system compliance (Experimental): effects of tidal volume guided by respiratory system compliance on mortality in patients suffering from ARDS
  Interventions: Behavioral: tidal volume guided by respiratory system compliance
- low tidal volume (Experimental): Ventilated patients with low tidal volume
  Interventions: Behavioral: low tidal volume

INTERVENTIONS:
Behavioral: tidal volume guided by respiratory system compliance — ventilated with tidal volume guided by respiratory system compliance
  Arms: tidal volume guided by respiratory system compliance
Behavioral: low tidal volume — ventilation ventilated with low tidal volume
  Arms: low tidal volume

SUMMARY:
The Acute Respiratory Distress Syndrome (ARDS) is one of common clinical critically diseases. In the United States, the incidence of ARDS reaches 31%, which is one of the main causes of death in patients. There is no unified treatment process for ARDS currently and the treatment measures are not yet standardized, so the standardization of ARDS treatment processes is needed to reduce mortality in patients. Following the evidence-based medicine principles and six-step treatment standards of ARDS, this study uses the method of multi-center randomized controlled clinical trials to evaluate the standardized treatment process of ARDS, which provides the basis for the standardized treatment of ARDS.

DETAILED DESCRIPTION:
From September 1st 2012 to September 30th 2014, all ARDS patients admitted to the ICUs will be enrolled. The demographic characteristics, diagnosis, formerly medical history, Ventilator indications, Ventilator data, other respiratory treatments, weaning outcome and 28 day mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years
2. admitted to the ICU
3. according to the diagnostic criteria of ARDS Berlin definition，admit patients with severe ARDS

Exclusion Criteria:

1. age <18 years old
2. be expected to die within 24 hours
3. end-stage malignancies
4. be participating in other studies, which may affect the results of this study
5. DNI (do not intubation) and DNR (do not recovery) patients
6. family members do not agree to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the effects of tidal volume guided by respiratory system compliance on mortality in patients suffering from ARDS | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Prof., Study Director — southeast university
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided